CLINICAL TRIAL: NCT02659488
Title: Effect of Lisdexamfetamine on Prefrontal Brain Dysfunction in Binge Eating Disorder
Brief Title: Lisdexamfetamine in Binge Eating Disorder (BED): fMRI Effects
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lindner Center of HOPE (Other)
Collaborators: University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2015-2882
Record Dates: First submitted 2016-01-08; First posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Binge Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lisdexamfetamine (Other): During the Treatment Phase, subjects will be evaluated after 1, 2, 3, 4, 6, 8, 10, and 12 weeks (see Figure 2). The morning after completing the first fMRI scan, LDX will be started at 30 mg q AM (Baseline). After 1 week, LDX will then be increased to 50 mg q AM (Visit 1); after another week, LDX will be increased to 70 mg q AM (Visit 2). A single downward dose titration to 50 mg is allowed during week 3 if 70 mg/d is not tolerated. LDX dose at week 4 (50 or 70 mg/d) will be maintained for the next 8 weeks. Patients who do not tolerate 50 or 70 mg/day will be terminated. For patients who complete the 12-week treatment phase, LDX will be stopped at week 12 visit.
  Interventions: Drug: Lisdexamfetamine

INTERVENTIONS:
Drug: Lisdexamfetamine — 20 healthy controls and 20 women subjects with BED agreeing to a 12-week, open-label trial of LDX and fMRI assessments immediately before and after the 12 weeks of LDX treatment will be recruited
  Other Names: Vyvanse

SUMMARY:
The purpose of this study is to explore the effect of Lisdexamfetamine on Prefrontal Brain Dysfunction in Binge Eating Disorder

DETAILED DESCRIPTION:
12-week, open-label LDX trial for BED including fMRI assessments to test the following specific predictions:

1. At baseline, patients with BED will show greater ventral prefrontal, striatal, and amygdala brain activation to high-calorie food pictures (reward) than matched healthy comparison subjects.
2. After 12 weeks of LDX treatment, BED will exhibit reduced ventral prefrontal, striatal and amygdala brain activation to food cues compared to baseline.
3. BED patients who display cessation of binge eating and those who demonstrate clinical improvement after 12 weeks of LDX treatment will show greater reductions in ventral prefrontal, striatal, and amygdala brain activation to food pictures than patients who do not stop binge eating and those who do not improve, respectively.

ELIGIBILITY:
Inclusion Criteria: Criteria for entering this study will include all of the following:

1. Subjects will meet the DSM-IV-TR criteria for a diagnosis of binge eating disorder (BED) for at least the last 6 months.
2. Subjects will report at least 3 binge eating (BE) days per week for the two weeks prior to LDX initiation prospectively documented in take-home binge diaries.
3. Women, through the ages of 18 and 55 years, inclusive.
4. Willingness to receive open-label LDX treatment for 12 weeks.
5. Willingness to receive an fMRI before and after 12 weeks of LDX treatment.

Exclusion Criteria:

Criteria for exclusion from this study will include all of the following:

1. Have concurrent symptoms of bulimia nervosa or anorexia nervosa.
2. Women who are pregnant, lactating, or of childbearing potential who are not using adequate contraceptive measures. The following are considered to be adequate methods of birth control: 1. intrauterine device (IUD); 2. barrier protection; 3. a contraceptive implantation system (Norplant); 4. oral contraceptive pills; 5. a surgically sterile patient; and 6. abstinence. All female subjects will have a negative pregnancy test prior to randomization.
3. Subjects who are displaying suicidal ideation on the Columbia-Suicide Severity Scale (C-SSRS) (21), or a suicide attempt within the last year as defined by the C-SSRS, or homicidality.
4. Subjects who are receiving a psychological (e.g., supportive psychotherapy, cognitive behavior therapy, interpersonal therapy) or weight loss (e.g., Weight Watchers) intervention for BED that was begun within the 3 months before study entry. Subjects who are receiving psychotherapy that was initiated prior to 3 months of the beginning of the study will be allowed to continue to receive their psychotherapy during the trial only if they agree to not make any changes to the frequency or nature of their psychotherapy during the course of the drug trial.
5. A DSM-IV-TR diagnosis of substance abuse or dependence (except nicotine abuse or dependence) within the 6 months prior to randomization.
6. Subjects who have used psychostimulants to facilitate fasting or dieting as a part of their eating disorder within the past 6 months; patients who have misused psychostimulants within the past 6 months; and patients who have a drug screen at the screening visit positive for psychostimulants.
7. A lifetime DSM-IV-TR history of ADHD, psychosis, mania or hypomania, or dementia.
8. History of any psychiatric disorder which might interfere with a diagnostic assessment, treatment, or compliance, or a current Montgomery Asberg Depression Scale (MADRS) (22) score ≥ 18.
9. Clinically unstable medical disease, including cardiovascular, hepatic, renal, gastrointestinal, pulmonary, metabolic, endocrine or other systemic disease; clinically significant abnormalities on physical exam; or clinically significant laboratory abnormalities. Subjects should be biochemically euthyroid to enter the study.
10. Have a history of a structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormality, coronary artery disease, stroke, or other serious cardiovascular problem.
11. History of seizures, including clinically significant febrile seizures in childhood.
12. Have uncontrolled hypertension (>160/100) or tachycardia (heart rate >110). m. Have an ECG with significant arrhythmias or conduction abnormalities, which in the opinion of the physician investigator preclude study participation.
13. Have clinically relevant abnormal laboratory results, specifically including hypokalemia.
14. Have a specific medical condition where LDX use is contraindicated, such as narrow angle glaucoma or Tourette's syndrome.
15. Subjects requiring treatment with any drug which might interact adversely with or obscure the action of the study medication. This includes warfarin, anticonvulsants, clonidine, theophylline, and pseudoephedrine.
16. Subjects who have received any psychotropic medications (other than hypnotics) within two weeks prior to LDX initiation, including monoamine oxidase inhibitors, tricyclics, selective serotonin reuptake inhibitors, antipsychotics, mood stabilizers, or psychostimulants.
17. Subjects who have received investigational medications or depot neuroleptics within three months prior to LDX initiation.
18. Subjects who have a known allergy to LDX or its constituents
19. An MRI scan is contraindicated in the subject for safety reasons, claustrophobia, or if the patient exceeds the weight limit of MRI scanner, ~350 pounds.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of ventral prefrontal, striatal, and amygdala brain activation, assessed using food cues. | Change from baseline to 12 weeks of brain activation
  Investigators will statistically compare the brain response to food pictures of BED patients before and after receiving 12 weeks of LDX treatment.

SECONDARY OUTCOMES:
Clinical Global Impression Improvement Scale (CGI-I) | weeks 1, 2, 3, 4, 6, 8, 10, 12
  score between 1-7 (1 = very much improved, ranging to 7 = very much worse)
Yale Brown Obsessive-Compulsive Scale modified for binge eating (YBOC-BE) | weeks 0,1, 2, 3, 4, 6, 8, 10, 12
  Will examine to see if severity of YBOC-BE scores correlate with fMRI abnormalities at baseline; and whether improvement in this scale with LDX treatment correlate with improvement in fMRI abnormalities at Endpoint.
Binge Eating Scale (BES) | weeks 0,1, 2, 3, 4, 6, 8, 10, 12
  Will examine to see if severity of BES scores correlate with fMRI abnormalities at baseline; and whether improvement in this scale with LDX treatment correlate with improvement in fMRI abnormalities at Endpoint.
Weight | weeks 0,1, 2, 3, 4, 6, 8, 10, 12
  measured in kilograms

CONTACTS AND LOCATIONS:
Overall Officials: Susan L McEroy, MD, Principal Investigator — Lindner Center of HOPE
Locations (1):
- Lindner Center of HOPE, Mason, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Study will be published in a peer-reviewed journal